CLINICAL TRIAL: NCT02896452
Title: Astronaut Vision Issues and One Carbon Metabolism: Expanded Polymorphism Evaluation and Evaluation in a Potential Analog Population
Brief Title: Astronaut Vision Issues in a Ground Analog Population: Polycystic Ovary Syndrome
Acronym: PCOS
Status: Active, not recruiting | Type: Observational
Sponsor: National Aeronautics and Space Administration (Unknown)
Collaborators: University of Texas (Other); Mayo Clinic (Other); University of Florida (Other); University of North Carolina (Other); Coastal Eye Associates (Unknown)
Responsible Party: Principal Investigator, Scott M. Smith, Nutritionist, Manager for Nutritional Biochemistry, National Aeronautics and Space Administration (NASA)
Organization: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Other Study IDs: NASA
Record Dates: First submitted 2016-08-24; First posted 2016-09-12 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Polycystic Ovarian Syndrome; Idiopathic Intracranial Hypertension
MeSH Terms: conditions — Polycystic Ovary Syndrome; Pseudotumor Cerebri

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The Mayo Clinic/NASA would like to keep the samples for future research. The subjects can still take part in the current study even if they don't want their sample to be used for future research. If the subject agrees to give their sample it will become the property of NASA. Some future studies may examine the DNA. The PI would contact the subject if there are findings which would be useful for the subjects' health care. The subject would be given general information on the potential risks, benefits, and costs of choosing to learn about the findings.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Women diagnosed with PCOS without IIH: Women diagnosed with polycystic ovary syndrome without idiopathic intracranial hypertension
- Women diagnosed with PCOS and IIH: Women diagnosed with polycystic ovary syndrome and idiopathic intracranial hypertension
- Women diagnosed with IIH without PCOS: Women diagnosed with idiopathic intracranial hypertension without polycystic ovary syndrome
- Women without PCOS or IIH: Women age and body mass index match controls without polycystic ovary syndrome or intracranial hypertension

SUMMARY:
The investigators have documented a genetic predisposition for some astronauts to develop ophthalmologic issues (e.g., choroidal folds, cotton wool spots, optic disc edema). Women with polycystic ovary syndrome (PCOS) have several characteristics similar to those described in astronauts, including: higher homocysteine concentrations, increased incidence of intracranial hypertension, increased retinal nerve fiber layer thickness, increased incidence of white matter hyperintensities on MRI, increased androgen concentrations (or androgen responses to space flight), and indices of altered carbohydrate metabolism. Women with PCOS have not been evaluated in detail regarding the occurrence of other anomalies observed in astronauts including choroidal folds, optic disc edema and cotton wool spots as well as changes in cycloplegic refraction, and optic nerve sheath diameter. While researchers have evaluated one-carbon metabolism pathway polymorphisms re: PCOS, and initial studies show an association with certain one-carbon polymorphisms, none have looked at the complete set of SNPs proposed here. This study will evaluate women with PCOS and/or idiopathic intracranial hypertension (IIH) to assess one-carbon biochemistry and genetics and their possible correlation with ophthalmologic findings. The investigators aim to clarify the relationship of one carbon metabolism and ophthalmic findings in astronauts and patients with PCOS and/or IIH.

DETAILED DESCRIPTION:
Evidence from initial analysis of 5 SNPs in the one-carbon metabolism pathway suggests that one-carbon pathway genes may predict risk of ocular changes and possible vision impairment during and after long-duration space flight. It is not precisely known whether it is these particular genes, or a haplotype of genes that are linked to these genes, that influence risk. Furthermore, ancestry is a strong factor that predicts SNP occurrence in a population, and the association between one-carbon metabolism and the risk of vision-related issues may simply stem from the fact that one particular ancestry has a higher prevalence of these SNPs.

The investigators propose that there are other SNPs in the one-carbon metabolism pathway that alter risk of ocular changes and potential vision impairment during long-duration spaceflight. To that end, extended studies of one-carbon genetics in astronauts have recently been initiated. The investigators hypothesize that the differences between genetic, biochemical, and ophthalmologic findings in PCOS and/or IIH patients and controls will mirror many of the differences found between astronauts who had ophthalmic issues during and after flight.

SPECIFIC AIMS

The key aims of this study are to: a) determine extensive one carbon pathway and related biochemistry, targeted metabolomics, and genetics (523 SNPs of the 85 major genes), and b) conduct ophthalmologic exams on patients in one of four treatment groups:

1. women diagnosed with PCOS without IIH
2. women diagnosed with PCOS and IIH
3. women diagnosed with IIH without PCOS
4. women without PCOS or IIH Participants will be matched by age and body mass index (BMI). Statistical analyses will be used to evaluate the independent and shared contributions of age, body mass (BMI), and genetics on biochemical, and ophthalmologic outcomes, with False Discovery Rate adjustments to account for multiple comparisons.

A secondary aim is to combine the patient and control data from this study with ISS crewmember data in order to help inform us on whether or not these two cohorts (astronauts with ophthalmic issues, PCOS patients) share similar associations among one-carbon metabolism genetics and biochemistry and ophthalmologic data identified in the investigators' earlier analyses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PCOS and/or IIH
* No current medications for the treatment of PCOS
* Age and BMI-matched healthy women without PCOS or IIH will be used as controls

Exclusion Criteria:

* Clinical diagnosis of Cushing's syndrome
* Untreated hypo/hyperthyroidism, elevated prolactin, congenital adrenal hyperplasia, renal insufficiency or diabetes.
* Currently taking medications that can affect androgen concentrations or insulin sensitivity.
* Pregnant, breast-feeding, taking oral contraceptives or currently smoking.
* Taking medications that affect folate or B12 metabolism, such as methotrexate, trimethoprim, triamterene, phenobarbital, phenytoin, carbamazepine, gabapentin, or primidone or topiramate.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Premenopausal women, age 18-50 years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Single Nucleotide Polymorphism (SNP) Genetic Testing related to 1-Carbon Metabolism Pathway for 523 SNPs | 1 Day
Ophthalmologic exam -OCT | 1 Day
  Optical coherence tomography test
Ophthalmologic exam -Fundus | 1 Day
  Fundus photography
Ophthalmologic exam - US | 1 Day
  Eye ultrasound exam
Ophthalmologic exam -Vision | 1 Day
  Cycloplegic refraction test
Ophthalmologic exam -IOP | 1 Day
  Intraocular pressure

SECONDARY OUTCOMES:
Questionnaire | 1 Day
  Questions related to birthplace, as well as birthplace of parents and grandparents, if known
B-vitamin Status - folate | 1 Day
  Serum Folate measurement
B-vitamin Status - B12 | 1 Day
  Methylmalonic acid
B-vitamin Status - serum B12 | 1 Day
  Serum vitamin B-12
Testosterone | 1 Day
Hemoglobin | 1 Day
Plasminogen Activator Inhibitor Antigen | 1 Day
Insulin | 1 Day
Homocysteine | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Smith, PhD, Principal Investigator — National Aeronautics and Space Administration (NASA); Alice Y Chang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon subject request.

REFERENCES:
- [Background] Zwart SR, Gregory JF, Zeisel SH, Gibson CR, Mader TH, Kinchen JM, Ueland PM, Ploutz-Snyder R, Heer MA, Smith SM. Genotype, B-vitamin status, and androgens affect spaceflight-induced ophthalmic changes. FASEB J. 2016 Jan;30(1):141-8. doi: 10.1096/fj.15-278457. Epub 2015 Aug 27. PMID 26316272
- [Background] Zwart SR, Gibson CR, Mader TH, Ericson K, Ploutz-Snyder R, Heer M, Smith SM. Vision changes after spaceflight are related to alterations in folate- and vitamin B-12-dependent one-carbon metabolism. J Nutr. 2012 Mar;142(3):427-31. doi: 10.3945/jn.111.154245. Epub 2012 Feb 1. PMID 22298570